CLINICAL TRIAL: NCT03004898
Title: Preventing Progression of Renal Disease by Multidisciplinary Education - A Cohort Study at Northern Taiwan.
Brief Title: Population-based Chronic Kidney Disease Cohort at Northern Taiwan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, I Wen Wu, MD, MD, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IWW-0006
Record Dates: First submitted 2016-10-14; First posted 2016-12-29 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Chronic Kidney Disease, Population, Community, Multidisciplinary, Education
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- education arm (Experimental): multidisciplinary education: multidisciplinary CKD education involving case management nurse, dietitian, social worker, pharmacists.
  Interventions: Behavioral: multidisciplinary renal education

INTERVENTIONS:
Behavioral: multidisciplinary renal education — multidisciplinary CKD care involving case management nurse, dietitian, social worker, pharmacists.

SUMMARY:
CKD is a global endemic disease with increased comorbidities and mortality. The prevalence and the incidence of the end-stage renal disease (ESRD) are extremely high in Taiwan. The prevalence of CKD remains high; however, the awareness remains low. Screening of unique risk factor and early diagnosis of CKD can improve outcome. Furthermore, data of renal education deep into the community remains limited. The aims of this study are:

1. Explore risk factors associated with CKD in the community
2. Establish multidisciplinary care model in the community
3. Investigate mechanistic mediators for CKD and multidisciplinary education approached in behavioral , physiological, immune and metabolomics aspects
4. Provide bio-specimen repository for future study

ELIGIBILITY:
Inclusion Criteria:

* residents of Northern Taiwan

Exclusion Criteria:

* pregnancy women, unwilling to participate

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2013-02; Primary Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
eGFR < 60 mL/min | through study completion, every 1 year
  change of renal function between groups
albuminuria/creatinine ratio >=30 | through study completion, every 1 year
  change of proteinuria between groups
proteinuria/creatine ratio >=150 | through study completion, every 1 year
  change of proteinuria between groups

SECONDARY OUTCOMES:
SF-36 | through study completion, every 1 year
  change of score between groups

CONTACTS AND LOCATIONS:
Overall Officials: I-Wen Wu, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Department of Nephrology, Chang Gung Memorial Hospital, Keelung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu IW, Wang SY, Hsu KH, Lee CC, Sun CY, Tsai CJ, Wu MS. Multidisciplinary predialysis education decreases the incidence of dialysis and reduces mortality--a controlled cohort study based on the NKF/DOQI guidelines. Nephrol Dial Transplant. 2009 Nov;24(11):3426-33. doi: 10.1093/ndt/gfp259. Epub 2009 Jun 2. PMID 19491379
- [Background] Chen SH, Tsai YF, Sun CY, Wu IW, Lee CC, Wu MS. The impact of self-management support on the progression of chronic kidney disease--a prospective randomized controlled trial. Nephrol Dial Transplant. 2011 Nov;26(11):3560-6. doi: 10.1093/ndt/gfr047. Epub 2011 Mar 17. PMID 21414969